CLINICAL TRIAL: NCT01119859
Title: A Multi-center, Randomized, Blinded, Parallel-group Study of the Reduction of Signs and Symptoms During Monotherapy Treatment With Tocilizumab 8 mg/kg Intravenously Versus Adalimumab 40 mg Subcutaneously in Patients With Rheumatoid Arthritis
Brief Title: A Study of Tocilizumab (RoActemra/Actemra) Versus Adalimumab in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA19924; 2009-015845-21
Record Dates: First submitted 2010-04-01; First posted 2010-05-10 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tocilizumab 8 mg/kg (Experimental): Patients received 6 infusions of tocilizumab 8 mg/kg intravenously every 4 weeks and 12 injections of placebo to adalimumab subcutaneously every 2 weeks.
  Interventions: Drug: Tocilizumab; Drug: Placebo to adalimumab
- Adalimumab 40 mg (Active Comparator): Patients received 12 injections of adalimumab 40 mg subcutaneously every 2 weeks and 6 infusions of placebo to tocilizumab intravenously every 4 weeks.
  Interventions: Drug: Adalimumab; Drug: Placebo to tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — The maximum dose was 800 mg for patients weighing more than 100 kg. Tocilizumab was infused into an arm vein over a 1-hour period.
  Other Names: RoActemra; Actemra
  Arms: Tocilizumab 8 mg/kg
Drug: Adalimumab
  Arms: Adalimumab 40 mg
Drug: Placebo to tocilizumab
  Arms: Adalimumab 40 mg
Drug: Placebo to adalimumab
  Arms: Tocilizumab 8 mg/kg

SUMMARY:
This randomized, blinded, parallel arm study evaluated the efficacy and safety of tocilizumab (RoActemra/Actemra) versus adalimumab as monotherapy in patients with rheumatoid arthritis who are intolerant of methotrexate or where continued treatment with methotrexate was considered inappropriate. Patients were randomized to receive either tocilizumab 8 mg/kg intravenously (iv) every 4 weeks plus placebo subcutaneously (sc) every 2 weeks, or adalimumab 40 mg sc every 2 weeks plus placebo iv every 4 weeks. Treatment was anticipated to last 24 weeks. With regard to the blind, the study nurse was unblinded due to the nature of the treatment administration, but the investigator and the patient remained blinded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age.
* Rheumatoid arthritis of > 6 months duration.
* Intolerant of methotrexate or continued treatment with methotrexate is considered inappropriate.
* All disease-modifying anti-rheumatic drugs (DMARD) are to be withdrawn prior to receiving study drug.
* Weight ≤ 150 kg.

Exclusion Criteria:

* Major surgery (including joint surgery) within 12 weeks prior to baseline or planned major surgery within 6 months after baseline.
* History of or current inflammatory joint disease other than rheumatoid arthritis (RA).
* Treatment with a biologic agent at any time prior to baseline.
* Intra-articular or parenteral corticosteroids ≤ 4 weeks prior to baseline.
* Active current infection or history of recurrent bacterial, viral, fungal or mycobacterial infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- United States (33):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - San Diego, California
  - Colorado Springs, Colorado
  - Trumbull, Connecticut
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Ormond Beach, Florida
  - Idaho Falls, Idaho
  - Springfield, Illinois
  - Cumberland, Maryland
  - Flowood, Mississippi
  - Tupelo, Mississippi
  - Lincoln, Nebraska
  - Dover, New Hampshire
  - New Brunswick, New Jersey
  - Hickory, North Carolina
  - Dayton, Ohio
  - Duncansville, Pennsylvania
  - Willow Grove, Pennsylvania
  - Wyomissing, Pennsylvania
  - Greenville, South Carolina
  - Hixson, Tennessee
  - Houston, Texas
  - Lubbock, Texas
  - Mesquite, Texas
  - Nassau Bay, Texas
  - Waco, Texas
  - Spokane, Washington
  - Tacoma, Washington
- Australia (2):
  - Maroochydore
  - Sydney
- Belgium (2):
  - Brussels
  - Liège
- Brazil (3):
  - Curitiba
  - Goiânia
  - São Paulo
- Prague, Czechia
- Finland (2):
  - Helsinki
  - Jyväskylä
- Germany (10):
  - Baden-Baden
  - Berlin
  - Cologne
  - Essen
  - Heidelberg
  - Herne
  - Hildesheim
  - Osnabrück
  - Ratingen
  - Würzburg
- Greece (3):
  - Athens
  - Heraklion
  - Thessaloniki
- Mexico (3):
  - Mexicali
  - Mexico City
  - Obregón
- Portugal (3):
  - Almada
  - Lisbon
  - Porto
- Spain (5):
  - A Coruña
  - Barcelona
  - Madrid
  - Santiago de Compostela
  - Seville
- Sweden (2):
  - Stockholm
  - Uppsala
- Switzerland (5):
  - Aarau
  - Geneva
  - Lausanne
  - Sankt Gallen
  - Zurich
- Turkey (Türkiye) (3):
  - Ankara
  - Antalya
  - Istanbul
- United Kingdom (5):
  - Cannock
  - Leeds
  - London
  - Newcastle upon Tyne
  - Poole

REFERENCES:
- [Derived] Strand V, Michalska M, Birchwood C, Pei J, Tuckwell K, Finch R, Gabay C, Kavanaugh A, Jones G. Impact of tocilizumab monotherapy on patient-reported outcomes in patients with rheumatoid arthritis from two randomised controlled trials. RMD Open. 2017 Sep 14;3(2):e000496. doi: 10.1136/rmdopen-2017-000496. eCollection 2017. PMID 28955499
- [Derived] Gabay C, McInnes IB, Kavanaugh A, Tuckwell K, Klearman M, Pulley J, Sattar N. Comparison of lipid and lipid-associated cardiovascular risk marker changes after treatment with tocilizumab or adalimumab in patients with rheumatoid arthritis. Ann Rheum Dis. 2016 Oct;75(10):1806-12. doi: 10.1136/annrheumdis-2015-207872. Epub 2015 Nov 27. PMID 26613768
- [Derived] Dennis G Jr, Holweg CT, Kummerfeld SK, Choy DF, Setiadi AF, Hackney JA, Haverty PM, Gilbert H, Lin WY, Diehl L, Fischer S, Song A, Musselman D, Klearman M, Gabay C, Kavanaugh A, Endres J, Fox DA, Martin F, Townsend MJ. Synovial phenotypes in rheumatoid arthritis correlate with response to biologic therapeutics. Arthritis Res Ther. 2014;16(2):R90. doi: 10.1186/ar4555. Epub 2014 Apr 30. PMID 25167216
- [Derived] Gabay C, Emery P, van Vollenhoven R, Dikranian A, Alten R, Pavelka K, Klearman M, Musselman D, Agarwal S, Green J, Kavanaugh A; ADACTA Study Investigators. Tocilizumab monotherapy versus adalimumab monotherapy for treatment of rheumatoid arthritis (ADACTA): a randomised, double-blind, controlled phase 4 trial. Lancet. 2013 May 4;381(9877):1541-50. doi: 10.1016/S0140-6736(13)60250-0. Epub 2013 Mar 18. PMID 23515142

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Started | 163 | 163
Completed | 139 | 133
Not Completed | 24 | 30
Not completed — Adverse Event | 9 | 10
Not completed — Death | 2 | 0
Not completed — Insufficient therapeutic response | 7 | 14
Not completed — Refused treatment | 3 | 6
Not completed — Failure to return | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg | Total
Number analyzed (Participants) | 163 | 162 | 325
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline Characteristics were analyzed for the intent-to-treat (ITT) population which included all randomized patients who received at least 1 dose of tocilizumab or adalimumab and had at least 1 efficacy assessment.
  One randomized patient in the adalimumab treatment group did not receive treatment and was not included in any of the data analyses, including demographics.
  years | 54.4 (12.95) | 53.3 (12.43) | 53.9 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristics were analyzed for the intent-to-treat (ITT) population which included all randomized patients who received at least 1 dose of tocilizumab or adalimumab and had at least 1 efficacy assessment.
  One randomized patient in the adalimumab treatment group did not receive treatment and was not included in any of the data analyses, including demographics.
  Participants
    Female | 129 | 133 | 262
    Male | 34 | 29 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in the Disease Activity Score 28 (DAS28)
Description: The DAS28 is a combined index for measuring disease activity in rheumatic arthritis (RA) and includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A negative change score indicates improvement. The analysis was adjusted for stratification factors of duration of RA (≤ 2 years and > 2 years) and region (US and non-US).
Time Frame: Baseline to Week 24
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of tocilizumab or adalimumab and had at least 1 efficacy assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Number analyzed (Participants) | 163 | 162
Units on a scale | -3.3 [-3.57 to -3.02] | -1.8 [-2.10 to -1.55]

2. Secondary Outcome: Percentage of Patients With a Remission Response (Disease Activity Score 28 [DAS28] < 2.6) at Week 24
Description: The percentage of patients who achieved remission of their rheumatic arthritis at Week 24, as measured by a DAS28 score < 2.6, is reported.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Number analyzed (Participants) | 163 | 162
Percentage of patients | 39.9 | 10.5

3. Secondary Outcome: Percentage of Patients With Low Disease Activity (Disease Activity Score 28 [DAS28] ≤ 3.2) at Week 24
Description: The percentage of patients who had low rheumatic arthritis disease activity at Week 24, as measured by a DAS28 score of 3.2 or less, is reported.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Number analyzed (Participants) | 163 | 162
Percentage of patients | 51.5 | 19.8

4. Secondary Outcome: Percentage of Patients With an Improvement of at Least 20%, 50%, or 70% in American College of Rheumatology (ACR) Score (ACR20/50/70) From Baseline at Week 24
Description: Improvement must be seen in tender and swollen joint counts (28 assessed joints) and in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, the extreme left end of the line "no disease activity" [symptom-free and no arthritis symptoms] and the extreme right end "maximum disease activity"; patient assessment of pain in previous the 24 hours on a VAS (extreme left end of the line "no pain" and the extreme right end "unbearable pain"); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and erythrocyte sedimentation rate.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Number analyzed (Participants) | 163 | 162
Percentage of patients
  ACR 20 response | 65.0 | 49.4
  ACR 50 response | 47.2 | 27.8
  ACR 70 response | 32.5 | 17.9

5. Secondary Outcome: Percentage of Patients With a European League Against Rheumatism (EULAR) Good Response at Week 24
Description: Change of the Disease Activity Score 28 score from baseline was used to determine EULAR responses of good, moderate, or no response. For a post-baseline score ≤ 3.2, a change from baseline of < -1.2 was a good response, < -0.6 to ≥ -1.2 was a moderate response, and ≥ -0.6 was no response. For a post-baseline score > 3.2 to ≤ 5.1, a change from baseline of < -0.6 was a moderate response and ≥ -0.6 was no response. For a post-baseline score > 5.1, a change from baseline < -1.2 was a moderate response and ≥ -1.2 was no response. A good response could not be achieved for post-baseline scores > 3.2.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Number analyzed (Participants) | 163 | 162
Percentage of patients | 51.5 | 19.8

6. Secondary Outcome: Percentage of Patients With a European League Against Rheumatism (EULAR) Good or Moderate Response at Week 24
Description: as for outcome 5
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Number analyzed (Participants) | 163 | 162
Percentage of patients | 77.9 | 54.9

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for each patient from Baseline until 12 weeks after the last infusion of a study treatment.
Description: Safety population: All patients who received at least 1 dose of tocilizumab or adalimumab and had at least 1 post-treatment safety assessment.
Arm/Group | Tocilizumab 8 mg/kg | Adalimumab 40 mg
Serious Adverse Events (participants affected / at risk) | 19/162 | 16/162
Other Adverse Events (participants affected / at risk) | 66/162 | 65/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=162) | Adalimumab 40 mg (N=162)
Cellulitis (Infections and infestations) | 0 | 2
Appendicitis perforated (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Infective tenosynovitis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral labyrinthitis (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=162) | Adalimumab 40 mg (N=162)
Upper respiratory tract infection (Infections and infestations) | 18 | 17
Nasopharyngitis (Infections and infestations) | 17 | 13
Urinary tract infection (Infections and infestations) | 9 | 11
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 9 | 15
Hypertension (Vascular disorders) | 13 | 7
Headache (Nervous system disorders) | 9 | 9
Nausea (Gastrointestinal disorders) | 6 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.